CLINICAL TRIAL: NCT04715256
Title: Interventional Study With Low Risks and Constraints on the Effect of KCNQ1 Mutation (Romano-Ward Syndrome) on Insulin Tolerance and Obsessive Compulsive Features, a Cross-sectional Study With Matched Controls With an Attempt of Linkage to Whole Genome Scanning.
Brief Title: Evaluation of the Effects of KCNQ1 Mutation on Insulin Tolerance and Obsessive Compulsive Features in Long QT Romano-Ward Syndrome Patients.
Acronym: PRIME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotrial (Industry)
Collaborators: European Union (Other); Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A02099-30; 847879 (Other Grant/Funding Number: European Union (Horizon 2020 program))
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Romano-Ward Syndrome; Long QT Syndrome; Compulsive Behavior; Healthy Individuals
Keywords: Romano-Ward Syndrome; Long QT Syndrome; Insulin-related diseases; Compulsive Behavior; ASBQ; CHIRP; OCI-R; UPPS-P; CPT; GWAS; Healthy individuals; KCNQ1 mutations
MeSH Terms: conditions — Romano-Ward Syndrome; Long QT Syndrome; Compulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KCNQ1 mutated subjects (Experimental): This arm includes :
  * KCNQ1-mutated subjects with long QT Romano-Ward syndrome
  * KCNQ1-mutated subjects without phenotypic expression of the Romano-Ward syndrome
  * family relatives of a KCNQ1-mutated enrolled subject, carrying the KCNQ1 family mutation
  Interventions: Behavioral: Cognitive assessment of obsessive-compulsive and impulsive behaviours; Genetic: Genomic analysis; Diagnostic Test: Glucoregulation assessment
- Healthy subjects (Sham Comparator): Healthy subjects will be matched to KCNQ1 subjects. The matching factors will be age per decade (18-28 years, > 28-38 years, > 38-48 years), gender and body mass index (BMI: ≤ 24.9 kg/m2; 25-29.9 kg/m2; > 30 kg/m2).
  Interventions: Behavioral: Cognitive assessment of obsessive-compulsive and impulsive behaviours; Genetic: Genomic analysis; Diagnostic Test: Glucoregulation assessment

INTERVENTIONS:
Behavioral: Cognitive assessment of obsessive-compulsive and impulsive behaviours — The content of the assessment will be the same for all subjects and will consist of a cognitive assessment (attention, impulsivity) and a clinical assessment (impulsive behaviour, autistic traits,obsessive-compulsive behaviour).
Genetic: Genomic analysis — A genome-wide association study (GWAS) will be performed for all subjects to search for associations between KCNQ1 mutations, insulin regulation and psychological features.
Diagnostic Test: Glucoregulation assessment — Fasted glycaemia and insulinaemia, glycated haemoglobin (HbA1c) and glycaemia following an oral glucose challenge test will be measured in all study subjects.

SUMMARY:
The objectives of the study are to investigate if KCNQ1 mutation in Romano-Ward long QT patients can be associated with changes in insulin regulation and with psychological features of compulsivity, impulsivity and behavioural rigidity.

DETAILED DESCRIPTION:
Romano-Ward Syndrome (RWS) is a rare disorder characterized by prolongation of the QT interval, as well as T-wave abnormalities and possibly polymorphic ventricular fibrillation. RWS is inherited in an autosomal dominant fashion. Mutations in the potassium voltage-gated channel subfamily Q Member 1 (KCNQ1), potassium voltage-gated channel subfamily H member 2 (KCNH2), sodium voltage-gated channel alpha subunit 5 (SCN5A), potassium voltage-gated channel subfamily E regulatory subunit 1 (KCNE1), and potassium voltage-gated channel subfamily E regulatory subunit 2 (KCNE2) genes are known to be causative, and these five genes together are responsible for virtually 100% of cases of RWS.

Dysregulation of insulin signalling has been implicated in multimorbidity across the lifespan, in particular in type 2 diabetes, metabolic syndrome, obesity and RWS. Numerous studies have shown a relationship between RWS and hyperinsulinemia. More recently, altered insulin signalling has also been implicated in neurodegenerative brain disorders, dementias and Alzheimer's disease. Diseases characterized by dysregulation of insulin signalling (i.e. insulinopathies) present a major health, societal, and economic burden. These insulin signalling-associated diseases are mostly chronic, and with limited or absent curative treatments. At the current time, the recognition and clinical management of insulin comorbidity remains poorly established; brain-based comorbidity is generally neglected, and medical efforts are only devoted to the management of the primary, somatic diagnosis.

The present study will be a part of the European Union (EU)-funded PRIME (for Prevention and Remediation of Insulin Multimorbidity in Europe) research program, which primary goal is to identify and specify the molecular mechanisms underlying the insulin multimorbidities through investigation of the diseases that cause the highest burden and costs to patients and society, and to outline new directions for research and clinical care thereof. The primary hypothesis of the PRIME project is that comorbidity observed in these somatic diseases (DM2, metabolic syndrome, obesity, RWS) is a result of dysregulated central and peripheral insulin signalling, downstream of synaptic dysfunction and of learning, memory, and executive functions impairments. This non-competitive EU Horizon2020 project will study the role of KCNQ1, a key molecule in insulin regulation, in the insulinopathies across different levels of organismal organisation.

The study will include 50 KCNQ1-mutated subjects (mainly RWS patients but also subjects carrying the KCNQ1 mutation but without phenotypic manifestation of long QT syndrome, and, because of the strong interest of the PRIME project in genetic analyses, family relatives carrying the same KCNQ1 mutation) and 50 matched healthy subjects. By comparing the test population to healthy subjects, the main objective of the trial is to test the hypothesis of an involvement of KCNQ1 in compulsivity, impulsivity and cognitive rigidity.

The insulin regulation evaluations will be performed by measuring glucose, insulin and glycated haemoglobin (HbA1c) in subjects. Compulsivity, impulsivity and behavioural rigidity will be assessed using 4 neuropsychological questionnaires (OCI-R, ASBQ, UPPS-P, CHIRP) and one objective test, the CPT.

Moreover, DNA extraction will be performed in order to search for associations between mutations, insulin regulation and psychological features in conducting a Genome-Wide Association Study (GWAS) (exploratory objective).

ELIGIBILITY:
Inclusion Criteria:

* In the investigator's opinion, the subject is generally healthy based on their medical records (subjects with KCNQ1 mutation only), medical history, physical examination, vital signs, body weight, ECG (except long QT if applicable), and based on the results of haematology, clinical chemistry, urinalysis, urine drug screen (UDS) and serology;
* Subjects with a KCNQ1 mutation: genotyped as having a mutation on the KCNQ1 gene with or without phenotypic manifestation of long QT syndrome;
* Relatives of subjects with a KCNQ1 mutation: KCNQ1-mutated family relatives (with or without phenotypic expression) of a subject carrying a KCNQ1 mutation (Romano-Ward patients or subjects without phenotypic manifestation of long QT syndrome);
* Relatives of subjects with a KCNQ1 mutation must live in a different household than the subject with the KCNQ1 mutation;
* All subjects: negative UDS by dipstick analysis: opiates, methadone, cocaine, amphetamines (including ecstasy), barbiturates, benzodiazepines, and cannabinoids at admission to the assessment visit;
* All subjects: negative alcohol breath test at admission to the assessment visit.

Exclusion Criteria:

* All subjects: having taken within 1 year before the assessment visit or currently taking any of the following medications: a. Antidiabetics: metformin, pioglitazone, acarbose, miglitol, sitagliptin, vildagliptin, saxagliptin, exenatide, liraglutide, semaglutide, repaglinide, nateglinide, insulin. b. Medications interfering with the central nervous system (CNS) such as any antipsychotic, antidepressant or regular use of anxiolytic medications > once a week, or any attention deficit/hyperactivity disorder (ADHD) medication (e.g. methylphenidate);
* Healthy subjects and relatives of subjects with a KCNQ1 mutation not phenotypically affected: any of the following on a de novo ECG: a. Heart rate (HR) < 40 bpm or > 100 bpm; b. PR interval <120 msec; c. Abnormal repolarization; d. QT interval corrected for HR using Fridericia's formula (QTcF) > 450 msec for male subjects or > 470 msec for female subjects.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Outcome related to glucoregulation : fasted glycemia | 15 minutes
  Plasma glucose concentration
Outcome related to glucoregulation : fasted insulin levels | 15 minutes
  Plasma insulin concentration
Outcome related to glucoregulation : glycated haemoglobin (HbA1c) | 15 minutes
  Blood HbA1c concentration
Outcome related to glucoregulation : glycemia 2hours following an oral glucose challenge | 2 hours
  Plasma glucose concentration

SECONDARY OUTCOMES:
Obsessive Compulsive Inventory-Revised (OCI-R) questionnaire total score and subscale scores | 30 minutes
  Subscales of OCI-R: washing, obsessing, hoarding, ordering, checking, neutralising
Adult Social Behaviour Questionnaire (ASBQ) total score and subscale scores | 30 minutes
  Subscales of ASBQ : reduced contacts, reduced empathy, reduced interpersonal insight, violations of social conventions, insistence of sameness, sensory stimulation and motor stereotypies.
Urgency, Premeditation, Perseverance, Sensation seeking, and Positive urgency scale (UPPS-P) subscale scores | 30 minutes
  Subscales of UPPS-P: negative urgency, lack of premeditation, lack of perseverance, sensation-seeking, positive urgency
Childhood Retrospective Perfectionism Questionnaire (CHIRP) total score | 30 minutes
  Total score
Continuous Performance Task (CPT) | 1 hour
  Variables of the CPT : omission errors, commission errors/false alarms, hits, hit rate, hit reaction time, difference between hit rate and false alarms rate (d').

OTHER OUTCOMES:
Genomic analyses (GWAS) | 15 minutes
  DNA methylation status at the KCNQ1 locus and Polygenic Risk Scores (PRS)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Hays, MD, Principal Investigator — Biotrial; Probst Vincent, MD, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - L'Institut du Thorax, Nantes Hospital, Nantes
  - Biotrial Clinical Unit, Rennes

IPD SHARING:
Plan to Share IPD: Yes
All anonymized individual participant data will be shared within the PRIME consortium collaborators in accordance with the PRIME Consortium Agreement
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data will be available starting in january 2023 and until december 2025

REFERENCES:
- [Background] Torekov SS, Iepsen E, Christiansen M, Linneberg A, Pedersen O, Holst JJ, Kanters JK, Hansen T. KCNQ1 long QT syndrome patients have hyperinsulinemia and symptomatic hypoglycemia. Diabetes. 2014 Apr;63(4):1315-25. doi: 10.2337/db13-1454. Epub 2013 Dec 18. PMID 24357532
- [Background] van de Vondervoort I, Poelmans G, Aschrafi A, Pauls DL, Buitelaar JK, Glennon JC, Franke B. An integrated molecular landscape implicates the regulation of dendritic spine formation through insulin-related signalling in obsessive-compulsive disorder. J Psychiatry Neurosci. 2016 Jun;41(4):280-5. doi: 10.1503/jpn.140327. PMID 26854754
- [Background] van de Vondervoort IIGM, Amiri H, Bruchhage MMK, Oomen CA, Rustogi N, Cooper JD, van Asten JJA, Heerschap A, Bahn S, Williams SCR, Buitelaar JK, Poelmans G, Glennon JC. Converging evidence points towards a role of insulin signaling in regulating compulsive behavior. Transl Psychiatry. 2019 Sep 12;9(1):225. doi: 10.1038/s41398-019-0559-6. PMID 31515486
- [Background] Southgate L, Tchanturia K, Collier D, Treasure J. The development of the childhood retrospective perfectionism questionnaire (CHIRP) in an eating disorder sample. Eur Eat Disord Rev. 2008 Nov;16(6):451-62. doi: 10.1002/erv.870. PMID 18444228
- [Background] Foa EB, Huppert JD, Leiberg S, Langner R, Kichic R, Hajcak G, Salkovskis PM. The Obsessive-Compulsive Inventory: development and validation of a short version. Psychol Assess. 2002 Dec;14(4):485-96. PMID 12501574
- [Background] Lynam, D.R., Smith, G.T., Whiteside, S.P., Cyders, M.A. (2006). The UPPS-P: Assessing five personality pathways to impulsive behavior (Technical Report). West Lafayette: Purdue University.
- [Background] Zermatten, A., Van der Linden, M., Jermann, F., Ceschi, G. Validation of a French version of the Obsessive-Compulsive Inventory-Revised in a non-clinical sample. (2006). Revue Européenne de Psychologie Appliquée. 56:151-155
- [Background] Van der Linden, M., d'Acremont, M., Zermatten, A., Jermann, F., Laroi, F., Willems, S., Juillerat, A., Bechara, A. (2006). A French Adaptation of the UPPS Impulsive Behavior Scale: Confirmatory factor analysis in a sample of undergraduate students. Eur J Psychol Assess. 22:38-42.
- [Result] Fatima SS, Chaudhry B, Khan TA, Farooq S. KCNQ1 rs2237895 polymorphism is associated with Gestational Diabetes in Pakistani Women. Pak J Med Sci. 2016 Nov-Dec;32(6):1380-1385. doi: 10.12669/pjms.326.11052. PMID 28083030
- See also: Official website of the PRIME project — https://prime-study.eu/
- See also: Biotrial's website — https://www.biotrial.com/